CLINICAL TRIAL: NCT05200975
Title: Pharmacokinetic and Pharmacodynamic Target Attainment of Cefuroxime in Adult Patients on General Wards With Different Degrees of Renal Function: a Prospective Observational Cohort Study
Brief Title: Target Attainment of Cefuroxim
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Noordwest Ziekenhuisgroep (Other)
Responsible Party: Principal Investigator, Saskia E. Zieck, Coordinating investigor, Noordwest Ziekenhuisgroep
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL78342.029.21
Record Dates: First submitted 2021-12-20; First posted 2022-01-21 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Infection, Bacterial; Kinesics
Keywords: cefuroxim; renal function; target attainment; infectious disease
MeSH Terms: conditions — Bacterial Infections; Kinesics; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Percentage of patients attaining the cefuroxime PK-PD target of 50%T>MIC. This will be investigated for patients with adequate renal function receiving a regular cefuroxime dose and impaired renal function receiving a guideline recommended reduced dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adequate renal function (Other): Patients with adequate renal function (egfr>30ml/min) receiving a regular cefuroxime dose
  Interventions: Diagnostic Test: Venapunction
- Impaired renal function (Other): Patients with impaired renal function (egfr<30ml/min) receiving a guideline recommended reduced dose
  Interventions: Diagnostic Test: Venapunction

INTERVENTIONS:
Diagnostic Test: Venapunction — Three venapunctures within a period of 72 hours, containing a maximum of 18ml of venous blood in total.

SUMMARY:
SUMMARY Rationale: Optimal antibiotic dosing in patients with bacterial infections is of high importance. Underdosing can lead to treatment failure and can promote emergence of antimicrobial resistance, while overdosing may lead to (harmful) side effects. The antibiotic cefuroxime is a second-generation cephalosporin and is frequently used in hospitalized patients. Cefuroxime exhibits, like other cephalosporins, time-dependent killing. The pharmacodynamic target can therefore be best described as the percentage of the dosing interval that the serum concentration remains above the minimum inhibitory concentration (MIC) of the bacteria (T>MIC). Attaining the pharmacokinetic-pharmacodynamic (PK-PD) target of 50%T>MIC is associated with antimicrobial therapeutic efficacy of cefuroxime.

Because cefuroxime is almost exclusively excreted through the kidneys, dose reduction of cefuroxime for patients with renal impairment (eGFR<30ml/min/1.73m2) is standard of care. No prospective evidence exists that currently guideline-recommended cefuroxime dosing regimens result in at least 50%T>MIC in adult patients on general wards, especially not in patients with renal impairment receiving a reduced dose of cefuroxime.

Objective: To investigate whether the PK-PD target of cefuroxime (50%T>MIC) is attained in the first 24 hours of treatment in adult patients on general wards with adequate and impaired renal function receiving regular and reduced doses of cefuroxime. Study design: Observational, prospective single center cohort study Study population: Adult patients (age ≥ 18 years) on general wards of Noordwest Ziekenhuisgroep (NWZ) receiving cefuroxime as part of standard care.

Intervention: Three venapunctures within a period of 72 hours, containing a maximum of 18ml of venous blood in total.

Main study parameters: Percentage of patients attaining the cefuroxime PK-PD target of 50%T>MIC. This will be investigated for patients with adequate renal function receiving a regular cefuroxime dose and impaired renal function receiving a guideline recommended reduced dose.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Risks imposed by participation are considered negligible. Three venapunctures, obtaining a maximum of 18 ml venous blood are not expected to cause AEs or SAEs. Participation itself does not bring any benefit as cefuroxime treatment is part of standard care, but the group related benefit could be significant. With the results of this study, current recommended cefuroxime dosing regimens are prospectively validated or an advice to reconsider current guidelines will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Receiving cefuroxime therapy intravenous (iv) as part of standard care
* Age ≥ 18 years
* Admitted to a general ward of Noordwest Ziekenhuisgroep - location Alkmaar
* Informed consent is obtained

Exclusion Criteria:

* Mentally incapacitated patients, i.e. a minor or legally incompetent adult
* Renal replacement therapy during treatment with cefuroxime
* Patients admitted to the intensive care unit (ICU)
* Severely burned patients, defined as a burned surface ≥ 10%
* Patients with cystic fibrosis
* Informed consent is not obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Target Attainment | 0-24hours after treatment initiation
  Main study parameter is the percentage of the study population attaining the target of 50%T>MIC within the first 24hrs of treatment. To calculate this endpoint cefuroxime concentrations and MIC-values will be obtained.

SECONDARY OUTCOMES:
Target Attainment | 0-48hours after treatment initiation
  Secondary study parameter is the percentage of the study population attaining the target of 50%T>MIC within the first 48hrs of treatment. To calculate this endpoint cefuroxime concentrations and MIC-values will be obtained.

CONTACTS AND LOCATIONS:
Locations (1):
- Noordwest Ziekenhuisgroep, Alkmaar, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided